CLINICAL TRIAL: NCT07263815
Title: EQUIP - Evaluation of Quality of Imaging on a Next-generation Total Body Pet Scan in Comparison to Conventional PET
Acronym: EQUIP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PMC121005 (25/150)
Record Dates: First submitted 2025-11-13; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: Total Body PET; EQUIP; Diagnostic; Imaging
MeSH Terms: conditions — Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging on Total Body PET (Experimental): Participants in this arm undergo a total body PET scan after conventional standard-of-care imaging
  Interventions: Device: PET

INTERVENTIONS:
Device: PET — This device images the whole body simultaneously with greater sensitivity allowing imaging to occur faster and with less radiation dose compared to conventional PET systems

SUMMARY:
The GE Healthcare Omni Total Body (TB) 128cms (Omni TB) is a long-axial field-of-view (LAFOV) PET/CT scanner and will be installed in a pre-market phase at the Peter MacCallum Cancer Centre.

The main features and functionality of this new scanner include high sensitivity, high resolution digital detectors based on silicon photomultipliers. The ultra-high sensitivity and extended field of view are designed to support the ability to reduce administrated dose and/or shorten acquisition time without compromising the image quality of the PET imaging.

To verify the appearance of images acquired on the Omni TB with images acquired on our conventional PET/CT equipment, a study imaging a cohort of patients on both devices is proposed. The study involves no additional radiopharmaceutical administration.

Additionally, in keeping with ALARA (as low as reasonably achievable) radiation dose practices, it will be possible to model acquisition settings (duration, administered activity and reconstruction parameters) using the system raw data and a suite of research tools to optimise acquisition parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, who is at least 18 years of age
2. Referred for a clinically indicated PET/CT scan with radiotracers F-18 FDG, F-18 DCFPyL, Ga-68 PSMA, Ga-68 DOTATATE or I-124
3. Able and willing to provide informed consent for participation in this study

Exclusion Criteria:

1) Known to be pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-11-24 (Estimated); Primary Completion 2026-02-24 (Estimated); Study Completion 2026-12-24 (Estimated)

PRIMARY OUTCOMES:
To assess the diagnostic quality of images acquired on the OMNI 128 Total Body PET | 1 Day
  To analyse the diagnostic image quality visually on the Omni TB with radiotracers F-18 FDG, F-18 DCFPyL, Ga-68 PSMA, Ga-68 DOTATATE or I-124

SECONDARY OUTCOMES:
To compare diagnostic image quality on the Omni TB with an existing PET/CT device | 1 Day
  Three nuclear medicine specialists will qualitatively assess diagnostic image quality using the the 5-point Likert visual grading score. Reviewers will be blinded to the clinical indication, camera model and reconstruction parameters prior to scoring to remove potential bias by expert reviewers.
To compare the sharpness and conspicuity of images produced on the Omni TB with an existing PET/CT device | 1 Day
  Three nuclear medicine specialists will qualitatively assess the sharpness and conspicuity of images using the the 5-point Likert visual grading score. Reviewers will be blinded to the clinical indication, camera model and reconstruction parameters prior to scoring to remove potential bias by expert reviewers.
To compare the noise characteristics of images acquired using the Omni TB with an existing PET/CT device | 1 Day
  Three nuclear medicine specialists will qualitatively assess the noise characteristics of images using the the 5-point Likert visual grading score. Reviewers will be blinded to the clinical indication, camera model and reconstruction parameters prior to scoring to remove potential bias by expert reviewers
To compare the quantitative parameters of SUVmean and SUVmax in normal organs on the Omni TB with an existing PET/CT device | 1 Day
  One nuclear medicine physician will create a region of interest (ROI) around seven normal tissues (kidneys, liver, spleen, muscle, brain, blood pool, and normal lung) to calculate the SUVmean and SUVmax. This assessment will be conducted on all images acquired to allow a comparison between imaging systems
To quantitatively compare the noise characteristics (signal to noise) of images acquired using the Omni TB with an existing PET/CT device | 1 Day
  The signal to noise ratio (SNR) will be determined by selecting a volume-of-interest (14cm3) in a region of normal liver. The standard deviation and mean of SUV values within this area will be calculated and used to determine the coefficient of variance (COV) by dividing the SUV standard deviation by the SUVmean. The SNR will then be calculated as the reciprocal of the COV
To compare the quantitative parameters of SUVmean, SUVmax and SUVpeak in up to three candidate lesions visualised on the Omni TB and an existing PET/CT device | 1 Day
  One nuclear medicine physician will create a spherical 2 cm region of interest (ROI) around up to three candidate lesions to calculate the SUVmean and SUVmax. Target lesion uptake will be determined by placing a 40% isocontour volume of interest (VOI) around the lesion and calculating SUVpeak. This assessment will be conducted on all images acquired to allow a comparison between imaging devices
To compare the visibility of lesions in images acquired using the Omni TB with images acquired on an existing PET/CT device | 1 Day
  To quantify the contrast between lesions and surrounding normal tissue the tumour to background ratio will be calculated as a function of the lesion SUVpeak over the SUV in the background. These values will be compared across imaging devices
To evaluate the quality of images obtained by the Omni TB with reduced scan time | 1 Day
  Patients imaged using the Omni TB system will have their images acquired for 10 minutes using LIST mode. This raw list mode data will be retrospectively reconstructed so only data over a specified time frame can be evaluated. Time frames will include, 10, 5, 2 and 1 min. These reconstructions will be analysed according to the secondary outcome measures 2 to 8
To evaluate the quality of images obtained by the Omni TB with reduced injected radioactivity | 1 Day
  Patients imaged using the Omni TB system will have their images acquired for 10 minutes using LIST mode. This raw list mode data will be retrospectively reconstructed to match the time per bed step used for the conventional PET/CT device. To simulate a lowered injection dose the LIST mode data will undergo Poisson resampling using the following factors, 1/2, 1/4, 1/8, 1/16

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hofman, Prof, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No